CLINICAL TRIAL: NCT04208893
Title: Combined Facility and Home-based Exercise Intervention of Supervised Aerobic Versus Combined Aerobic and Strength Training in Children With Repaired Tetralogy of Fallot: A Feasibility Pilot Trial
Brief Title: Exercise Training Strategies for Children With Repaired Tetralogy of Fallot
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study suspended due to COVID-19 restrictions.
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian McCrindle, Staff Cardiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000062584
Record Dates: First submitted 2019-11-08; First posted 2019-12-23 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Tetralogy of Fallot; Congenital Heart Defects; Congenital Abnormalities; Cardiovascular Diseases; Heart Diseases
Keywords: Pediatrics; Tetralogy of Fallot; Exercise intervention; Physical fitness; Congenital Heart Defects; Exercise rehabilitation
MeSH Terms: conditions — Tetralogy of Fallot; Heart Defects, Congenital; Congenital Abnormalities; Cardiovascular Diseases; Heart Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic training only (Experimental): The aerobic training intervention will include 60 minutes/session, 3 times/week for 12 weeks at an intensity of 65% - 85% of participants' heart rate reserve (HRR), as determined by the CPET. Patients will be asked to wear a fitness-tracking device to monitor their heart rate response and in order to comply with the prescribed training intensity. All training sessions will start with a 10-minute warm up, 40-minute aerobic interventions, and ends with 10-minute of cool down. One study doctor will be on call during in-hospital training. Onsite supervised aerobic interventions will include play-based activities, whereas home-based aerobic activities will include stationary bikes and exercise activities that would target desired heart rate ranges. Home exercise equipment will be provided.
  Interventions: Behavioral: Exercise training
- Combined aerobic and strength training (Experimental): Participants in this group will perform a combination of aerobic and strength training activities for 60 minutes/session, 3 times/week for 12 weeks. Aerobic activities for this group will be similar to Arm 1. Strength training will be based on participant's individual assessment findings and developmental status. Resistance level will be set at approximately 50% of the patient maximal load and increased by 3 pounds (or the next level of resistance band) once the patient is able to perform 30 repetitions. Closed kinetic chain exercises such as pushups, squats, and lunges will be made more challenging by the addition of weight or change in body position. Training sessions will include a 10-minute warm up, 40-minute aerobic and strength exercises, and a 10-minute cooldown.
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — See description of Arms

SUMMARY:
The investigators will explore the feasibility and safety of two exercise interventions delivered both in the hospital and in participants' homes. Preteens and adolescents who have had repaired Tetralogy of Fallot (TOF), will be grouped by age and randomly assigned to either an aerobic or strength training exercise program supervised for 12 weeks. An exploratory aim of this study will be to examine changes in fitness level, muscle strength, muscle oxygen extraction and quality of life after the intervention, and compare these measures between groups. At the end of the study, participants and parents will be interviewed to assess their satisfaction and ideas for improvements in the program.

DETAILED DESCRIPTION:
While adult cardiac rehabilitation (CR) is an established clinical practice, the conceptualization, design and utility of pediatric CR programs have been poorly studied. Particular challenges for children with heart disease include uncertainties regarding physical activity restrictions imposed by clinicians and overprotection by caregivers. These challenges may lead to poor lifestyle and deconditioning, resulting in increased health risks associated with inactivity, such as adiposity, and reduced perceived general health and quality of life. Preliminary studies have shown therapeutic benefits of physical exercise as an add-on therapy in an effort to improve patients' functional outcome after cardiac surgery 1; however, delivery of these programs has been variable, and it is not clear whether a combined program of facility and home-based exercise would yield higher patient adherence for children. The investigators hypothesize that a supervised exercise training program delivered both in the hospital and in participants' homes will be acceptable and feasible for children with repaired Tetralogy of Fallot (TOF). The investigators will conduct a pilot trial over 1 year in which the investigators will randomize 20 participants to either aerobic exercise only or a combined aerobic and strength training program for 12 weeks. The investigators will conduct qualitative interviews to understand intervention acceptability. Results will support a larger definitive study aimed at determining efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls ages 10 to 17 years with repaired Tetralogy of Fallot, currently followed at The Hospital for Sick Children, Toronto, Ontario
* Participant fluent in English

Exclusion Criteria:

* Moderate-to-severe ventricular dysfunction at the latest echocardiogram (defined as the qualitative grade given on the echocardiogram done closest to the intervention)
* Previous history of or documented frequent premature atrial or ventricular contractions or runs or associated tachycardia at the latest exercise test
* Reside outside 50km radius from SickKids or >1hour travel distance to SickKids
* Lack of internet and computer/laptop access
* Skeletal muscle or orthopedic pathologies
* Neurodevelopmental delay that would preclude participation in an exercise program
* History of syncope with exercise
* Planned surgery requiring admission to intensive care unit during the study intervention

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Consent rate | 1 year
  The proportion of participants consented to participate in the study
Enrolment rate | 1 year
  The proportion of participants who consented and eligible to participate in the study
Adherence rate | 1 year
  The proportion of participants who adhered to the study intervention based on the number of completed training sessions divided by the total number of training sessions available
Completion rate | 1 year
  The proportion of participants who completed the study intervention
Attrition rate | 1 year
  The proportion of participants who withdrew or lost to follow up
Acceptability questionnaire (Investigator-generated satisfaction questionnaire) | 1 year
  The proportion of participants who were satisfied with the study intervention. An investigator-generated satisfaction questionnaire was created to assess the many components of acceptability of the exercise intervention program. Participants will be provided with statements related to the study intervention, for example "the exercises were enjoyable", and participant will rate these statements based on whether they Strongly Agree, Agree, Neither Agree nor Disagree, Disagree, and Strongly Disagree

SECONDARY OUTCOMES:
7. The effect of aerobic training only versus combined aerobic and strength training on exercise capacity using cardiopulmonary exercise test in children with repaired Tetralogy of Fallot (TOF) (peak exercise ml/kg/min) | From baseline to 3 months post intervention
  Change in time in oxygen consumption at peak exercise (ml/kg/min). The cardiopulmonary exercise test will be used report objective values for oxygen consumption at peak exercise.
The effect of aerobic training only versus combined aerobic and strength training on pulmonary measures using pulmonary function test in children with repaired Tetralogy of Fallot (TOF) (Change in time in force vital capacity (FVC) (liters)) | From baseline to 3 months post intervention
  Change in time in force vital capacity (FVC) (liters)
The effect of aerobic training only versus combined aerobic and strength training on pulmonary measures using pulmonary function test in children with repaired Tetralogy of Fallot (TOF) (Change in time in predicted force vital capacity (FVC) (liters)) | From baseline to 3 months post intervention
  Change in time in predicted force vital capacity (FVC) (liters)
The effect of aerobic training only versus combined aerobic and strength training on pulmonary measures using pulmonary function test in children with repaired Tetralogy of Fallot (TOF) (Change in time in percent predicted force vital capacity (FVC) (%)) | From baseline to 3 months post intervention
  Change in time in percent predicted force vital capacity (FVC) (%)
The effect of aerobic training only versus combined aerobic and strength training on pulmonary measures using pulmonary function test in children with repaired Tetralogy of Fallot (TOF) Change in time forced expiratory volume within one second (FEV1) (L) | From baseline to 3 months post intervention
  Change in time in forced expiratory volume within one second (FEV1) (liters)
The effect of aerobic training only versus combined aerobic and strength training on pulmonary measures using pulmonary function test in children with repaired Tetralogy of Fallot (TOF) Change in time predicted Forced expiratory volume (FEV1) (L) | From baseline to 3 months post intervention
  Change in time in predicted Forced expiratory volume (FEV1) (liters)
The effect of aerobic training only versus combined aerobic and strength training on pulmonary measures using pulmonary function test in children with repaired Tetralogy of Fallot (TOF) Change in time percent predicted Forced expiratory volume (FEV1) | From baseline to 3 months post intervention
  Change in time in percent predicted Forced expiratory volume (FEV1) (%)
The effect of aerobic training only versus combined aerobic and strength training on pulmonary measures using pulmonary function test in children with repaired Tetralogy of Fallot (TOF) (Change in time in FEV1/FVC (%)) | From baseline to 3 months post intervention
  Change in time in FEV1/FVC (%)
The effect of aerobic training only versus combined aerobic and strength training on pulmonary measures using pulmonary function test in children with repaired Tetralogy of Fallot (TOF) (Change in time in predicted FEV1/FVC (%)) | From baseline to 3 months post intervention
  Change in time in predicted FEV1/FVC (%)
The effect of aerobic training only versus combined aerobic and strength training on pulmonary measures using pulmonary function test in children with repaired Tetralogy of Fallot (TOF) (Change in time in maximum voluntary ventilation (MVV) (L/min)) | From baseline to 3 months post intervention
  Change in time in maximum voluntary ventilation (MVV) (L/min)
The effect of aerobic training only versus combined aerobic and strength training on pulmonary measures using pulmonary function test in children with repaired Tetralogy of Fallot (TOF) Change in time in predicted Max voluntary ventilation (MVV) (L/min) | From baseline to 3 months post intervention
  Change in time in predicted Maximum voluntary ventilation (MVV) (L/min)
The effect of aerobic training only versus combined aerobic and strength training on pulmonary measures using pulmonary function test in children with repaired Tetralogy of Fallot (TOF) Change in time in % predicted Max voluntary ventilation (MVV) | From baseline to 3 months post intervention
  Change in time in percent predicted Maximum voluntary ventilation (MVV) (%)
The effect of aerobic training only versus combined aerobic and strength training on muscle strength using a handheld dynamometer (JAMAR) in children with repaired Tetralogy of Fallot (TOF) | From baseline to 3 months post intervention
  Change in time in grip strength (kg)
The effect of aerobic training only versus combined aerobic and strength training on flexibility using the sit-and-reach test in children with repaired Tetralogy of Fallot (TOF) | From baseline to 3 months post intervention
  Change in time in flexibility of the lower back and hamstring muscles (cm)
The effect of aerobic training only versus combined aerobic and strength training on muscle strength using the Bruininks-Oseretsky Test of Motor Proficiency-2 (BOT-2) in children with repaired Tetralogy of Fallot (TOF) | From baseline to 3 months post intervention
  Change in time in running speed agility (scale score from 1-30, higher score mean better outcome)
The effect of aerobic training only versus combined aerobic and strength training on running speed and agility using the Bruininks-Oseretsky Test of Motor Proficiency-2 (BOT-2) in children with repaired Tetralogy of Fallot (TOF) | From baseline to 3 months post intervention
  Change in time in muscle strength (scale score from 1-30, higher score mean better outcome)
The effect of aerobic training only versus combined aerobic and strength training on participant-reported quality of life (QoL) questionnaire score in children with repaired Tetralogy of Fallot (TOF) | From baseline to 3 months post intervention
  Change in participant-reported QoL questionnaire (PedsQL 4.0: Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales). The self-reported QoL questionnaire PedsQL 4.0 is composed of 23 items comprising 4 dimensions. Each item is rated with a 5-point Likert response scale from 0 to 4 (0=never, 1=almost never, 2=sometimes, 3=often, and 4=almost always). Items are reversed scored and linearly transformed to a 0-100 scale. Higher scores indicate better quality of life
The effect of aerobic training only versus combined aerobic and strength training on parent-reported quality of life (QoL) questionnaire score in children with repaired Tetralogy of Fallot (TOF) | From baseline to 3 months post intervention
  Change in parent-reported QoL questionnaire (PedsQL 4.0: Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales). The parent-reported QoL questionnaire PedsQL 4.0 is composed of 23 items comprising 4 dimensions. Each item is rated with a 5-point Likert response scale from 0 to 4 (0=never, 1=almost never, 2=sometimes, 3=often, and 4=almost always). Items are reversed scored and linearly transformed to a 0-100 scale. Higher scores indicate better quality of life
The effect of aerobic training only versus combined aerobic and strength training on participant-reported quality of life (QoL) questionnaire score (PedsQLTM 3.0 Cardiac Module) in children with repaired Tetralogy of Fallot (TOF) | From baseline to 3 months post intervention
  Change in participant-reported QoL questionnaire (PedsQLTM 3.0 Cardiac Module). The self-reported PedsQLTM 3.0 Cardiac Module is composed of 23 items comprising 6 dimensions. Each item is rated with a 5-point Likert response scale from 0 to 4 (0=never, 1=almost never, 2=sometimes, 3=often, and 4=almost always). Items are reversed scored and linearly transformed to a 0-100 scale. Higher scores indicate lower problem.
The effect of aerobic training only versus combined aerobic and strength training on parent-reported quality of life (QoL) questionnaire score (PedsQLTM 3.0 Cardiac Module) in children with repaired Tetralogy of Fallot (TOF) | From baseline to 3 months post intervention
  Change in parent-reported QoL questionnaire (PedsQLTM 3.0 Cardiac Module). The parent-reported PedsQLTM 3.0 Cardiac Module is composed of 23 items comprising 6 dimensions. Each item is rated with a 5-point Likert response scale from 0 to 4 (0=never, 1=almost never, 2=sometimes, 3=often, and 4=almost always). Items are reversed scored and linearly transformed to a 0-100 scale. Higher scores indicate lower problem.
The effect of aerobic training only versus combined aerobic and strength training on participant-reported quality of life (QoL) questionnaire score (PedsQLTM Multidimensional Fatigue Scale) in children with repaired Tetralogy of Fallot (TOF) | From baseline to 3 months post intervention
  Change in participant-reported QoL questionnaire (PedsQLTM Multidimensional Fatigue Scale). The self-reported PedsQLTM Multidimensional Fatigue Scale is composed of 18 items comprising 3 dimensions. Each item is rated with a 5-point Likert response scale from 0 to 4 (0=never, 1=almost never, 2=sometimes, 3=often, and 4=almost always). Items are reversed scored and linearly transformed to a 0-100 scale. Higher scores indicate lower problem.
The effect of aerobic training only versus combined aerobic and strength training on parent-reported quality of life (QoL) questionnaire score (PedsQLTM Multidimensional Fatigue Scale) in children with repaired Tetralogy of Fallot (TOF) | From baseline to 3 months post intervention
  Change in parent-reported QoL questionnaire (PedsQLTM Multidimensional Fatigue Scale). The parent-reported PedsQLTM Multidimensional Fatigue Scale is composed of 18 items comprising 3 dimensions. Each item is rated with a 5-point Likert response scale from 0 to 4 (0=never, 1=almost never, 2=sometimes, 3=often, and 4=almost always). Items are reversed scored and linearly transformed to a 0-100 scale. Higher scores indicate lower problem.
The effect of aerobic training only versus combined aerobic and strength training on muscle Tissue Saturation Index (TSI) using near-infrared spectroscopy device after Tetralogy of Fallot (TOF) repair | From baseline to 3 months post intervention
  Change in time in muscle Tissue Saturation Index (TSI) (%)
The effect of aerobic training only versus combined aerobic and strength training on muscle oxygenation using near-infrared spectroscopy device after Tetralogy of Fallot (TOF) | From baseline to 3 months post intervention
  Change in time in muscle oxygenation (O2Hb) (%)
The effect of aerobic training only versus combined aerobic and strength training on muscle deoxygenation using near-infrared spectroscopy device after Tetralogy of Fallot (TOF) repair | From baseline to 3 months post intervention
  Change in time in muscle deoxygenation (HHb) (%)
The effect of aerobic training only versus combined aerobic and strength training on muscle morphology using ultrasound imaging after Tetralogy of Fallot (TOF) repair | From baseline to 3 months post intervention
  Change in time in quadriceps muscles thickness (cm)
The effect of aerobic training only versus combined aerobic and strength training on anthropometric measures in children with repaired Tetralogy of Fallot (TOF) (Change in time in body mass index (kg/m^2)) | From baseline to 3 months post intervention
  Change in time in body mass index (kg/m^2)
The effect of aerobic training only versus combined aerobic and strength training on anthropometric measures in children with repaired Tetralogy of Fallot (TOF) (Change in time in waist circumference (cm)) | From baseline to 3 months post intervention
  Change in time in waist circumference (cm)
The effect of aerobic training only versus combined aerobic and strength training on anthropometric measures in children with repaired Tetralogy of Fallot (TOF) (Change in time in waist/height ratio (WHtR)) | From baseline to 3 months post intervention
  Change in time in waist/height ratio (WHtR)
The effect of aerobic training only versus combined aerobic and strength training on self-efficacy participation to physical activity after Tetralogy of Fallot (TOF) repair | From baseline to 3 months post intervention
  Change in time in Children's Self-perceptions of Adequacy and Predilection for Physical Activity (CSAPPA) scale. CSAPPA is a 20-item scale designed to capture children's perceived adequacy to perform physical activities and preference to either physical activity engagement or sedentary pursuit. It is composed of 3 subscales related to physical activity: adequacy (7 items), predilection (9 items), and enjoyment of physical education class (3 items). Each item was structured in an alternative choice format whereby children will be asked to select an option that best describes them. For example, children will choose which of these two statements best identify them "some kids can't wait to play active games after school" or "other kids would rather do something else", then indicate whether the selected claim was either "sort of true for me" or "really true for me". Each response is scored from 1 to 4, where highest score indicate preference to more active endeavours.
The effect of aerobic training only versus combined aerobic and strength training on participant's readiness to change behaviour after Tetralogy of Fallot (TOF) repair | From baseline to 3 months post intervention
  Change in time in readiness to change score. the Readiness to Change questionnaire is based on the Transtheoretical Stages of Change Model where an individual's motivation to change behaviour, in the context of exercise/physical activity participation, is classified into 1 of the 5 stages of change which are precontemplation, contemplation, preparation, action, and maintenance.
8. The effect of aerobic training only versus combined aerobic and strength training on exercise capacity using cardiopulmonary exercise test in children with repaired Tetralogy of Fallot (TOF) (anerobic exercise ml/kg/min) | From baseline to 3 months post intervention
  Change in time in oxygen consumption at anaerobic exercise (ml/kg/min). The cardiopulmonary exercise test will be used report objective values for oxygen consumption at anaerobic exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Brian McCrindle, MD, Principal Investigator — The Hospital for Sick Children, Toronto, Canada
Locations (1):
- Brian W. McCrindle, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Williams CA, Wadey C, Pieles G, Stuart G, Taylor RS, Long L. Physical activity interventions for people with congenital heart disease. Cochrane Database Syst Rev. 2020 Oct 28;10(10):CD013400. doi: 10.1002/14651858.CD013400.pub2. PMID 33112424